CLINICAL TRIAL: NCT02742883
Title: A Phase 2 Study of Atengenal (A-10) and Astugenal (AS2-1) in Diffuse, Intrinsic Pontine Glioma (DIPG)
Brief Title: A Study of Atengenal and Astugenal in Diffuse, Intrinsic Pontine Glioma (DIPG)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical Hold
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI-BT-55
Record Dates: First submitted 2016-04-12; First posted 2016-04-19 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Diffuse, Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for up to 104 days. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dosage is reached, but not exceeding 12.0 g/kg/d Atengenal or 0.4 mg/kg/d Astugenal.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with diffuse intrinsic pontine glioma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for diffuse, intrinsic pontine glioma (DIPG) provide very limited benefit to the patient. The rationale for the use of Antineoplaston therapy in this protocol study derives from experience with subjects from prior Phase 2 studies and Compassionate Exemption patients treated with Antineoplaston therapy at the Burzynski Clinic.

This study is designed to analyze the efficacy and safety of Antineoplaston therapy in five separate DIPG patient cohorts, which are defined by age and prior therapy. This is a two stage study with 20 patients in each cohort being enrolled in the first stage and an additional 20 patients being enrolled in the second stage, if pre-determined efficacy endpoints in the first stage are realized.

DETAILED DESCRIPTION:
This study is designed to analyze the response of diffuse, intrinsic brainstem glioma (DIPG) to Antineoplaston therapy in 5 separate patient cohorts, which are defined by age and prior therapy. The primary endpoint is objective response (OR), but the determination of OR in DIPG is problematic. Determination of OR using the Macdonald, RANO, and RECIST criteria relies on postgadolinium TI-weighted MRI images of enhancing disease. However, DIPG shows variable enhancement and has a non-enhancing component as seen on T2/FLAIR-weighted MRI images. Recent reviews have proposed OR assessment in diffuse low grade gliomas using modified RANO criteria and in recurrent glioblastoma using RECIST + F (T2/FLAIR-weighted images).Neither of these methodologies have been validated.

This single-arm Phase 2 study of the efficacy of Antineoplaston therapy in DIPG will utilize both bidimensional assessment of enhancing DIPG (RANO), a validated primary endpoint, and unidimensional assessment of enhancing + non-enhancing DIPG (RECIST + F), an exploratory endpoint.

This Phase 2 protocol has a strategy for early assessment of response rates with procedures for termination of enrollment for lack of efficacy. A minimax two-stage design is utilized.

Ten patients with enhancing disease will be enrolled in stage 1 for each cohort. If none of the 10 patients in a particular cohort achieves an OR based on bidimensional measurements, no additional patients with enhancing disease will be enrolled into that particular cohort. However, if 1 of the 10 patients with enhancing disease in a particular cohort achieves an OR, then an additional 10 patients with enhancing disease will be enrolled in stage 2 of the minimax design for that cohort, yielding a maximum of 20 patients with enhancing disease for that cohort. As exploratory endpoints, complete response (CR), partial response (PR), and progressive disease (PD) rates, as well as 6-, 12-, and 24-month overall survival (OS) will be analyzed.

Patients with no enhancing disease will also be enrolled into each cohort but will not count against the numbers designated in the two-stage minimax design. An exploratory endpoint for these patients will be 6-, 12-, and 24-month OS.

Other exploratory endpoints will be determination of OR, CR, PR, and PD based on unidimensional measurement of the enhancing + non-enhancing components of DIPG (RECIST + F).

At completion of this study, the efficacy of Antineoplaston therapy in each cohort and the desirability of its further development in any particular cohort will be determined in discussion with the FDA.

ELIGIBILITY:
Inclusion Criteria:

Five cohorts of patients with diffuse, intrinsic pontine glioma will be studied:

1. Patients age 3 months to < 3 years;
2. Patients age 3-21 years with progressive disease (PD) following radiation therapy (RT) ± chemotherapy and/or other therapies;
3. Patients age 3-21 years with newly diagnosed DIPG who (or whose parents / guardians) have refused RT;
4. Patients age > 21 years with PD following RT ± chemotherapy and/or other therapies; and
5. Patients age > 21 years with newly diagnosed DIPG who have refused RT.

Exclusion Criteria include:

1. Disseminated disease, multicentric tumors, or leptomeningeal disease;
2. Uncontrolled intercurrent illness;
3. A history of New York Heart Association Class II congestive heart failure or above;
4. Pregnancy.

Ages: 3 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy Measured by Objective Response Rate | 104 weeks
  Objective Response Rate

SECONDARY OUTCOMES:
Efficacy Measured by Overall Survival | 6 months, 12 months, and 24 months
  6 months, 12 months, and 24 months overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com